CLINICAL TRIAL: NCT03632239
Title: Reverse Phenotyping Core (RPC)
Brief Title: Reverse Phenotyping Core
Status: Enrolling by invitation | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 180129; 18-HG-0129
Record Dates: First submitted 2018-08-14; First posted 2018-08-15 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01-21

CONDITIONS: Harboring of Unexpected Genetic Variant
Keywords: Resource; Variant; Sequencing; Genome; Phenotype; Natural History

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Reverse Phenotyping Core: Individuals undergoing phenotyping by the Reverse Phenotyping Core (RPC)

SUMMARY:
Background:

Genes tell a person's body how to grow and work. All people have variations in their genes. Some of these cause differences that show up in a person's traits or their health, others do not. Researchers want to gather more data on people based on their genes. They want to use this data to learn more about diseases and possible treatments.

Objectives:

To develop a cohort of participants who can be contacted again for phenotyping and collect their genetic data. To share those data with other researchers and make them searchable.

Eligibility:

People already enrolled in a wide variety of protocols. They will be of varying health status, age, and sex. They will have had or plan to have exome or genome sequencing under their protocol. They can be re-contacted by the research team for possible other studies.

Design:

Participants will give basic details like contact and demographic information.

Participants may answer questions about their personal health history, their family medical history, or their thoughts or reactions to data.

Participants may have basic health tests. Their height, weight, or blood pressure may be checked.

Participants may have tests of heart function. They may have an ultrasound or other non-invasive test.

Participants may provide blood, urine, or other samples.

Participants may have scans or other tests.

Participants will get the results of all clinical tests in a letter.

If any tests are abnormal, someone from the study will call the participant to explain what the results mean and what to do about them.

Participants will get genetic testing results only if researchers think they could affect the health of the participant or their relatives.

DETAILED DESCRIPTION:
Study Design:

RPC will be a data resource of genetic variants with the capability of performing phenotyping for selected study participants who have undergone genome or exome sequencing and were consented for data sharing and re-contact. De-identified genome or exome data will be collected as the RPC Genomic Data Archive and available in a web browser quantifying alleles in aggregate. Investigators may request additional data for research on the basis of variants of interest identified in the browser. Individuals with genetic variants of interest may be offered phenotyping under RPC. Phenotyping performed under RPC will include obtaining medical information, gathering biologic samples, and selected diagnostic studies that can be performed in the NIHCC (NIH Clinical Center). RPC will enable investigation of phenotypic consequences of genetic variation in humans by using a genomic ascertainment strategy to minimize the bias of phenotypic ascertainment.

Primary Objective:

1. To pilot the development of a cohort of individuals with genome or exome sequencing data who can be re-contacted for phenotyping and make those data available to and searchable by collaborators.
2. To facilitate the completion of genotype-driven research projects by RPC or other investigators.

Secondary Objectives:

Secondary objectives will relate to the studies that will address phenotypic consequences of specific genetic variants identified in the RPC cohort. Such studies will include investigation of the phenotypic spectrum associated with genetic variation.

Endpoints:

This is a hypothesis-generating research study and therefore has no concrete endpoints.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participants in the RPC Genomic Data Archive must have exome or genome sequencing available that collaborators have permission to share for inclusion in our resource.
* Participants in the RPC Genomic Data Archive must be re-contactable by the primary study team (e.g., the collaborator who contributes their data must be able to contact the participants).
* All participants must be >= 4 years old.
* Health Perceptions Survey Criterion: Only adult participants who are able to provide consent for themselves will be eligible for this portion of the study.

Ages: 4 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals who have undergone genome sequencing under separate protocol
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-01-23 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-12-29 (Estimated)

PRIMARY OUTCOMES:
Hypotheses from RPC to be tested | yearly
  RPC will generate data regarding phenotypic consequences of genetic variants

CONTACTS AND LOCATIONS:
Overall Officials: Clesson E Turner, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
We are actively depositing data into the database of genotypes and phenotypes (dbGaP), which is designed with tiered access to clinical data. That is, there is open, public access to summary clinical data of study participants and qualified investigators may apply for access to individual, coded clinical results. Such access is limited to authorized medical researchers and redistribution and security policies are strict. Broad future use of the data deposited into dbGaP (as opposed to restricted use for specific disorders) will be permitted. Sequence traces for individual genes will be available publicly (deposited in GenBank); however, these sequence traces will not be linked to a participant's identifiable information, nor to the sequence traces of other genes sequenced in that participant's sample. Coded genomic data are available to data contributors and NIH intramural investigators through the Reverse Phenotyping Core browser (18-HG-0129; https://rpc.nhgri.nih.gov/).
Supporting Information: Study Protocol
Time Frame: Data in dbGap is stored per NIH policy. Data in the Reverse Phenotyping Core/TGAC browser will be stored for the remainder of the protocol (18-HG-0129) and the time the study is closed, a proposal to the IRB will be made to keep the data or destroy it.
Access Criteria: dbGap is a controlled-access database with view-only access to summary-level information and individual-level genotype and sequence data associated with phenotypic features. The Reverse Phenotyping Core/TGAC browser allows researchers to identify particular genotypes or ranges of genotypes, while preserving the privacy of study participants by only displaying aggregate data for one or a limited number of loci in a search. The browser is located on NIH servers and searchable only by investigators in the NIH s intramural research program or external collaborators who have contributed sequence data.

REFERENCES:
- [Background] Wilczewski CM, Obasohan J, Paschall JE, Zhang S, Singh S, Maxwell GL, Similuk M, Wolfsberg TG, Turner C, Biesecker LG, Katz AE. Genotype first: Clinical genomics research through a reverse phenotyping approach. Am J Hum Genet. 2023 Jan 5;110(1):3-12. doi: 10.1016/j.ajhg.2022.12.004. PMID 36608682
- [Background] Garnai SJ, Brinkmeier ML, Emery B, Aleman TS, Pyle LC, Veleva-Rotse B, Sisk RA, Rozsa FW, Ozel AB, Li JZ, Moroi SE, Archer SM, Lin CM, Sheskey S, Wiinikka-Buesser L, Eadie J, Urquhart JE, Black GCM, Othman MI, Boehnke M, Sullivan SA, Skuta GL, Pawar HS, Katz AE, Huryn LA, Hufnagel RB; Genomic Ascertainment Cohort; Camper SA, Richards JE, Prasov L. Variants in myelin regulatory factor (MYRF) cause autosomal dominant and syndromic nanophthalmos in humans and retinal degeneration in mice. PLoS Genet. 2019 May 2;15(5):e1008130. doi: 10.1371/journal.pgen.1008130. eCollection 2019 May. PMID 31048900
- [Background] Manthiram K, Preite S, Dedeoglu F, Demir S, Ozen S, Edwards KM, Lapidus S, Katz AE; Genomic Ascertainment Cohort; Feder HM Jr, Lawton M, Licameli GR, Wright PF, Le J, Barron KS, Ombrello AK, Barham B, Romeo T, Jones A, Srinivasalu H, Mudd PA, DeBiasi RL, Gul A, Marshall GS, Jones OY, Chandrasekharappa SC, Stepanovskiy Y, Ferguson PJ, Schwartzberg PL, Remmers EF, Kastner DL. Common genetic susceptibility loci link PFAPA syndrome, Behcet's disease, and recurrent aphthous stomatitis. Proc Natl Acad Sci U S A. 2020 Jun 23;117(25):14405-14411. doi: 10.1073/pnas.2002051117. Epub 2020 Jun 9. PMID 32518111
- [Background] Johnston JJ, Brennan ML, Radenbaugh B, Yoo SJ, Hernandez SM; NHGRI Reverse Phenotyping Core; Lewis KL, Katz AE, Manolio TA, Biesecker LG. The ACMG SF v3.0 gene list increases returnable variant detection by 22% when compared with v2.0 in the ClinSeq cohort. Genet Med. 2022 Mar;24(3):736-743. doi: 10.1016/j.gim.2021.11.012. Epub 2021 Nov 18. PMID 34906458
- [Background] Spontarelli K, Young VC, Sweazey R, Padro A, Lee J, Bueso T, Hernandez RM, Kim J, Katz A, Rossignol F, Turner C, Wilczewski CM, Maxwell GL, Holmgren M, Bailoo JD, Yano ST, Artigas P. ATP1A1-linked diseases require a malfunctioning protein product from one allele. Biochim Biophys Acta Mol Cell Res. 2024 Jan;1871(1):119572. doi: 10.1016/j.bbamcr.2023.119572. Epub 2023 Sep 1. PMID 37659504
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2018-HG-0129.html